CLINICAL TRIAL: NCT01099189
Title: A Cohort Study of the Histopathological Changes Evident in Vein Wall at the Time of Arteriovenous Dialysis Access Fistulas and the Effects of Such Changes on Biomechanical Compliance and Patient's Clinical Outcomes in a University Teaching Hospital.
Brief Title: Vein Histology in Arteriovenous Fistulas and Its Effect on Fistula Surgery Success
Status: Completed | Type: Observational
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Collaborators: University of Hull (Other)
Responsible Party: Sponsor
Other Study IDs: Access 4
Record Dates: First submitted 2010-04-05; First posted 2010-04-06 (Estimated); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Renal Replacement Therapy; Arteriovenous Fistula
Keywords: Histology; Compliance; Dialysis; Arteriovenous access fistula; vein
MeSH Terms: conditions — Arteriovenous Fistula; Patient Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — vein samples collected at time of fistula formation
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observed cohort: All patients recruited. Observed for clinical outcomes

SUMMARY:
Patients whose kidneys have failed need to receive dialysis treatment, most commonly with a dialysis machine. In order to be connected to the machine an operation is often performed to join an artery to a vein in the arm. This forms what is known as an arteriovenous fistula. The fistula causes an increase in the flow of blood through the vein and the vein reacts to this by becoming bigger and thicker, making it easier to connect the patient to the machine.

The success rate for the operation is relatively low and only approximately 65 from every 100 operations is still working after a year. It is thought that one factor that may cause problems with the fistula is the ability of the vein to stretch in response to increased blood flow. Previous research has shown that veins in kidney failure patients look different to those of people whose kidneys are working when viewed under a microscope.

The investigators aim to study the structure of the vein that is used in making fistulas with a microscope and also to test it in an engineering laboratory to see how much it will stretch. The investigators hope that gaining information about the structure of the vein and its ability to stretch will help determine what it is about the vein that affects how well it works as part of a fistula. This information may help surgeons select the best possible vein in a given patient to give the best chance of a working fistula in the future.

ELIGIBILITY:
Inclusion Criteria:

1. Patients referred to vascular consultants for AV fistula formation for haemodialysis access.
2. Ability to give informed written consent
3. Aged over 18 at time of referral

Exclusion Criteria:

1. Veins identified on preoperative ultrasound scanning to be of a calibre too small to allow sufficient material to be obtained for biomechanical testing (<3mm diameter).
2. Inability to give informed written consent
3. Aged under 18 at time of referral
4. Inability to attend follow-up appointments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patient referred for access formation
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2010-07; Primary Completion 2012-10 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Primary failure of access - Immediate/early thrombosis or failure to mature. | within 30 days of formation
  Failure to mature or thrombosis of fistula

SECONDARY OUTCOMES:
Duplex findings of evidence of stenosis and correlation to compliance or histological findings | 6 months
Correlation between biomechanical compliance and histological measures of pre existing venous pathology | 6 months
Correlation between biomechanical compliance testing and clinical outcomes | 6 months
Assisted primary and secondary patency rates at 3 and 6 months post fistula formation | 6 months
Functional primary patency | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ian C Chetter, MBChB FRCS, Principal Investigator — University of Hull
Locations (1):
- Academic Vascular Surgery Unit, Hull, Yorkshire, United Kingdom

REFERENCES:
- [Result] Smith GE, Gohil R, Chetter IC. Factors affecting the patency of arteriovenous fistulas for dialysis access. J Vasc Surg. 2012 Mar;55(3):849-55. doi: 10.1016/j.jvs.2011.07.095. Epub 2011 Nov 8. PMID 22070937